CLINICAL TRIAL: NCT00134004
Title: A Phase II Trial of Non-Myeloablative Conditioning and Transplantation of Partially HLA-Mismatched Bone Marrow for Patients With Hematologic Malignancies
Brief Title: Fludarabine, Cyclophosphamide, and Total-Body Irradiation in Treating Patients Who Are Undergoing a Donor Bone Marrow Transplant for Hematologic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J0457 CDR0000440990; P01CA015396 (NIH); P30CA006973 (NIH); JHOC-J0457 (Other: Johns Hopkins SKCCC); JHOC-04072704
Record Dates: First submitted 2005-08-22; First posted 2005-08-24 (Estimated); Results first posted 2015-08-24 (Estimated); Last update posted 2015-10-06 (Estimated); Status verified 2015-09

CONDITIONS: Chronic Myeloproliferative Disorders; Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes
Keywords: adult acute lymphoblastic leukemia in remission; adult acute myeloid leukemia in remission; childhood acute lymphoblastic leukemia in remission; childhood acute myeloid leukemia in remission; childhood chronic myelogenous leukemia; chronic phase chronic myelogenous leukemia; refractory chronic lymphocytic leukemia; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); chronic idiopathic myelofibrosis; chronic myelomonocytic leukemia; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; noncontiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II mantle cell lymphoma; noncontiguous stage II marginal zone lymphoma; noncontiguous stage II small lymphocytic lymphoma; recurrent adult Burkitt lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult Hodgkin lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent/refractory childhood Hodgkin lymphoma; recurrent childhood large cell lymphoma; recurrent childhood lymphoblastic lymphoma; recurrent childhood small noncleaved cell lymphoma; nodal marginal zone B-cell lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; refractory multiple myeloma; relapsing chronic myelogenous leukemia; secondary myelodysplastic syndromes; splenic marginal zone lymphoma; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; stage III adult Burkitt lymphoma; stage III adult diffuse large cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult Hodgkin lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III mantle cell lymphoma; stage III marginal zone lymphoma; polycythemia vera; essential thrombocythemia; stage III small lymphocytic lymphoma; stage IV mantle cell lymphoma; stage IV marginal zone lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV adult Burkitt lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV small lymphocytic lymphoma; stage IV adult Hodgkin lymphoma; childhood myelodysplastic syndromes
MeSH Terms: conditions — Myeloproliferative Disorders; Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Leukemia, Myeloid, Chronic-Phase; Leukemia, Lymphocytic, Chronic, B-Cell; Congenital Abnormalities; Primary Myelofibrosis; Leukemia, Myelomonocytic, Chronic; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Recurrence; Dendritic Cell Sarcoma, Interdigitating; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Polycythemia Vera; Thrombocythemia, Essential | interventions — Cyclophosphamide; fludarabine phosphate; Mycophenolic Acid; Tacrolimus; Radiotherapy

ARMS (1):
- Mini-haplo Transplant (Experimental): Non-myeloablative haploidentical bone marrow transplant with a fludarabine, cyclophosphamide (Cy), TBI (total body irradiation) preparative regimen and post-transplant Cy, mycophenolate mofetil (MMF), and tacrolimus as GVHD prophylaxis.
  Interventions: Drug: cyclophosphamide; Drug: fludarabine phosphate; Drug: mycophenolate mofetil; Drug: tacrolimus; Procedure: allogeneic bone marrow transplantation; Radiation: radiation therapy

INTERVENTIONS:
Drug: cyclophosphamide
Drug: fludarabine phosphate
Drug: mycophenolate mofetil
Drug: tacrolimus
Procedure: allogeneic bone marrow transplantation
Radiation: radiation therapy

SUMMARY:
RATIONALE: Giving low doses of chemotherapy, such as fludarabine and cyclophosphamide, and radiation therapy before a donor bone marrow transplant helps stop the growth of cancer cells. Giving chemotherapy or radiation therapy before or after transplant also stops the patient's immune system from rejecting the donor's bone marrow stem cells. The donated stem cells may replace the patient's immune system cells and help destroy any remaining cancer cells (graft-versus-tumor effect). Sometimes the transplanted cells from a donor can also make an immune response against the body's normal cells. Giving tacrolimus and mycophenolate mofetil after the transplant may stop this from happening.

PURPOSE: This phase II trial is studying how well giving fludarabine and cyclophosphamide together with total-body irradiation works in treating patients who are undergoing a donor bone marrow transplant for hematologic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine transplant-related mortality, risk of relapse, and progression-free survival of patients with standard- or high-risk hematologic malignancies undergoing nonmyeloablative conditioning comprising fludarabine, cyclophosphamide, and total-body irradiation followed by HLA-haploidentical allogeneic bone marrow transplantation.
* Determine donor hematopoietic chimerism in patients' peripheral blood at 30, 60, and 180 days after transplantation.
* Determine hematologic and nonhematologic toxic effects of this regimen in these patients.
* Determine, when feasible, surface expression of HLA molecules and death receptors, sensitivity to cytotoxic lymphocytes, and expression of anti-apoptotic genes (e.g., Bcl-2, Bcl-xL, X-IAP, and c-FLIP) in cancer cells from patients who relapse after treatment with this regimen.

OUTLINE: This is a multicenter study. Patients are stratified according to risk of relapse (standard [defined as ≤ 30% risk] vs high [defined as ≥ 70% risk]).

* Nonmyeloablative conditioning regimen: Patients receive fludarabine IV over 30 minutes on days -6 to -2 and cyclophosphamide IV over 1-2 hours on days -6 and -5. Patients undergo total body irradiation on day -1.
* Allogeneic bone marrow transplantation: Patients undergo donor bone marrow infusion on day 0.
* Post-transplantation therapy: Patients receive cyclophosphamide IV over 1-2 hours on days 3 and 4.
* Graft-vs-host disease prophylaxis: Beginning on day 5, patients receive oral mycophenolate mofetil 3 times daily until day 35 and tacrolimus IV (then changing to orally) twice daily until day 180.

Treatment continues in the absence of disease progression.

After completion of study transplantation, patients are followed on days 30, 60, 100, and 180; at 1 year; and then annually for 4 additional years.

PROJECTED ACCRUAL: A total of 75-100 patients will be accrued for this study within 3-4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of 1 of the following hematologic malignancies:

  * Acute leukemia

    * In second or subsequent complete remission (CR), as defined by absence of abnormal blast population by flow cytometry
    * In first CR with any of the following poor-risk cytogenetic features:

      * Alteration of chromosome 5 or 7
      * Multiple abnormalities
      * Philadelphia chromosome positive
  * Chronic phase chronic myelogenous leukemia (CML)

    * In first chronic phase and refractory to interferon alfa or imatinib mesylate
    * In second or subsequent chronic phase
  * Chronic lymphocytic leukemia, meeting 1 of the following criteria:

    * Received prior chemotherapy with a nucleoside analog and had remission lasting < 6 months
    * Received 1 prior therapy and has any of the following high-risk features:

      * Cytogenetic abnormalities of 17p, 11q
      * Mutations of the Zap70 gene
      * Somatically unmutated immunoglobulin heavy chain variable region genes
  * Hodgkin's lymphoma

    * Ineligible for autologous stem cell transplantation (SCT) due to any of the following exclusion factors:

      * LVEF < 45%
      * FEV_1 or FVC < 50% of predicted (75% of predicted in patients with prior thoracic or mantle radiotherapy)
      * Total bilirubin > 2.0 mg/dL (unless documented Gilbert's disease)
      * Creatinine > 2.0 mg/dL
  * Non-Hodgkin's lymphoma (NHL)

    * Low-grade NHL allowed provided patient had a remission duration of < 1 year after administration of any established, multi-agent chemotherapy regimen (e.g., CVP, CHOP, or rituximab in combination with CHOP)
    * Intermediate- or high-grade NHL allowed provided patient is ineligible for autologous SCT according to the criteria listed above
  * Multiple myeloma
  * Myelodysplastic syndromes
  * Paroxysmal nocturnal hemoglobinuria
  * Chronic myeloproliferative disorders other than CML, including any of the following:

    * Chronic myelomonocytic leukemia
    * Agnogenic myeloid metaplasia (or myeloid metaplasia with myelofibrosis), with hemoglobin < 10 g/dL OR WBC < 4,000/mm^3 or > 30,000/mm^3
    * Polycythemia vera or essential thrombocythemia in "spent" phase, with a history of 2 of the following:

      * Marrow fibrosis
      * Splenomegaly
      * Cytopenia (i.e., absolute neutrophil count < 1,500/mm^3, platelet count < 100,000/mm^3, hemoglobin < 10 g/dL)
    * Polycythemia vera or essential thrombocythemia with transformation to myelodysplastic syndromes or acute myeloid leukemia (requires treatment to achieve < 20% blasts in marrow)
* No smoldering myeloma
* Patients with acute myeloid leukemia or myelodysplastic syndromes must have had comprehensive cytogenetic evaluation of bone marrow specimen during active disease
* Ineligible for or refused bone marrow transplantation from an HLA-matched sibling or unrelated donor
* Ineligible for or refused autologous SCT
* Must have an HLA mismatched (i.e., 3/6, 4/6, or 5/6) related (first-degree relative)* donor available

  * Donor ≥ 18 years of age NOTE: *Patients with an inherited recombinant HLA haplotype may receive marrow from the parent in whose gamete the recombination occurred

NOTE: A new classification scheme for adult non-Hodgkin's lymphoma has been adopted by PDQ. The terminology of "indolent" or "aggressive" lymphoma will replace the former terminology of "low", "intermediate", or "high" grade lymphoma. However, this protocol uses the former terminology.

PATIENT CHARACTERISTICS:

Age

* 6 months to 74 years

Performance status

* ECOG 0-1

Life expectancy

* Not specified

Hematopoietic

* See Disease Characteristics

Hepatic

* See Disease Characteristics
* Bilirubin < 3.1 mg/dL

Renal

* See Disease Characteristics

Cardiovascular

* See Disease Characteristics
* LVEF ≥ 35%

Pulmonary

* See Disease Characteristics
* FEV_1 or FVC ≥ 40% of predicted in patients without prior thoracic or mantle radiotherapy (60% of predicted in patients with prior thoracic or mantle radiotherapy)

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* HIV negative
* Geographically accessible
* No debilitating medical or psychiatric illness that would preclude giving informed consent or receiving optimal treatment or follow-up

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Disease Characteristics
* No prior transfusions from donor

Chemotherapy

* See Disease Characteristics

Endocrine therapy

* Not specified

Radiotherapy

* See Disease Characteristics

Surgery

* Not specified

Ages: 6 Months to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2004-10; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ephraim J. Fuchs, MD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (3):
- United States (3):
  - Blood and Marrow Transplant Program at Northside Hospital, Atlanta, Georgia
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Hahnemann University Hospital, Philadelphia, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Groups:
- Mini-haplo BMT: Non-myeloablative haploidentical bone marrow transplant with a fludarabine, cyclophosphamide (Cy), TBI (total body irradiation) preparative regimen and post-transplant Cy, mycophenolate mofetil (MMF), and tacrolimus as GVHD prophylaxis.
Period: Overall Study
Arm/Group | Mini-haplo BMT
Started | 210
Completed | 210
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Mini-haplo BMT
Number analyzed (Participants) | 210
Age, Continuous [Mean (Full Range); unit: years] | 52 [1 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61
  Male | 149
Region of Enrollment [Number; unit: participants]
  United States | 210

OUTCOME MEASURES:

1. Primary Outcome: Transplant-related Mortality
Description: Percentage of participants who die for any reason other than recurrence of disease.
Time Frame: Cumulative incidence for the entire study, up to 11 years
Measure: Number; unit: percentage of participants
Arm/Group | Mini-haplo BMT
Number analyzed (Participants) | 210
percentage of participants | 18

2. Primary Outcome: Relapse Rate
Description: Percentage of participants who experience disease relapse.
Time Frame: Cumulative incidence for the entire study, up to 11 years
Measure: Number; unit: percentage of participants
Arm/Group | Mini-haplo BMT
Number analyzed (Participants) | 210
percentage of participants | 55

3. Primary Outcome: Progression-free Survival
Description: Percentage of participants who do not experience disease relapse, disease progression, or death.
Time Frame: 2 years
Measure: Number; unit: percentage of participants
Arm/Group | Mini-haplo BMT
Number analyzed (Participants) | 210
percentage of participants | 34

4. Secondary Outcome: Graft Failure Rate
Description: Percentage of participants who experienced failure to engraft (also called graft failure or graft rejection). Failure to engraft is defined as <5% donor chimerism and absence of relapse or any other reason for that chimerism value. All participants who met this criterion were included in this outcome measure.
Time Frame: Cumulative incidence for the entire study, up to 11 years
Measure: Number; unit: percentage of participants
Arm/Group | Mini-haplo BMT
Number analyzed (Participants) | 210
percentage of participants | 13

5. Secondary Outcome: Hematologic and Non-hematologic Toxicities as Measured by NCI Common Toxicity Criteria for Adverse Events, v 3.0 Weekly Until 1 Year After Transplantation
Description: Percentage of study participants who experienced a serious adverse event (SAE) within 1 year of bone marrow transplant. Complete data is provided in the Adverse Event tables.
Time Frame: 1 year
Measure: Number; unit: percentage of participants
Arm/Group | Mini-haplo BMT
Number analyzed (Participants) | 210
percentage of participants | 9.5

ADVERSE EVENTS:
Arm/Group | Mini-haplo BMT
Serious Adverse Events (participants affected / at risk) | 20/210
Other Adverse Events (participants affected / at risk) | 11/210
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mini-haplo BMT (N=210)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 2 (2)
Altered mental status (Nervous system disorders) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1)
Cholestasis (Gastrointestinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fungemia (Infections and infestations) | 3 (3)
GI bleed (Gastrointestinal disorders) | 2 (2)
Idiopathic pneumonia syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Multi-organ failure (Investigations) | 1 (1)
Neutropenic fever (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 5 (5)
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 1 (1)
Pulmonary Vascular Obstructive Disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 4 (4)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 8 (8)
Seizure (Nervous system disorders) | 1 (1)
Sepsis (Infections and infestations) | 6 (6)
Subdural hematoma (Vascular disorders) | 3 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mini-haplo BMT (N=210)
Pneumonia (Infections and infestations) | 11 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No